CLINICAL TRIAL: NCT04586075
Title: UW Undiagnosed Genetic Diseases Program
Status: Recruiting | Type: Observational
Sponsor: University of Wisconsin, Madison (Other)
Collaborators: University of Wisconsin Center for Human Genomics and Precision Medicine (Unknown)
Responsible Party: Sponsor
Other Study IDs: 2020-0700; SMPH (Other: UW Madison); Protocol Version 10/28/2024 (Other: UW Madison)
Record Dates: First submitted 2020-10-06; First posted 2020-10-14 (Actual); Last update posted 2025-06-04 (Actual); Status verified 2025-05

CONDITIONS: Rare Diseases; Genetic Disease; Undiagnosed Disease
Keywords: genomics; genome sequencing; undiagnosed disease
MeSH Terms: conditions — Rare Diseases; Genetic Diseases, Inborn; Undiagnosed Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood samples will be collected on all probands, parents, and participating affected family members unless they are refused by the participant or their collection would compromise participant safety. For a minority of patients, other biological samples may also be requested i.e., urine collection, saliva/buccal smears, and punch skin biopsies. Samples whose collection involves more than minimal risk (i.e., cerebrospinal fluid, bone marrow, liver, muscle, conjunctival, or renal biopsy) will be opportunistically obtained from residual material left after procedures performed for clinical purposes.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Undiagnosed Disease Group: Blood or other relevant biological samples obtained from consenting research subjects will be banked and extracted for DNA and RNA.
  Interventions: Diagnostic Test: Trio Whole Genome Sequencing and Participant-Specific Research

INTERVENTIONS:
Diagnostic Test: Trio Whole Genome Sequencing and Participant-Specific Research — The initial evaluation begins with short-read genome sequencing of DNA extracted from blood of affected individual(s) and participating family members (The most common approach will be trio whole genome sequencing, which involves the affected child + their parents).
  Additional evaluation may include: functional assessments, animal modeling, reverse phenotyping (may require an interim visit), epigenetic profiling, or clinical database matching through selective sharing of coded patient data with external collaborators (e.g., via Matchmaker Exchange and Phenome Central), long read genome sequencing, de novo genome assembly, RNA sequencing, and novel bioinformatics analyses

SUMMARY:
The primary purpose of this study is to discover new disease genes for rare Mendelian disorders and its secondary purpose include diagnosing people with rare genetic disorders that have not been previously diagnosed through conventional clinical means, learning more about the pathobiology of genetic disorders, and developing novel diagnostic technologies and analytics. 500 participants with undiagnosed and suspected genetic disorders will be recruited.

DETAILED DESCRIPTION:
An estimated 10,000 rare Mendelian genetic disorders affect, in aggregate, one in twelve individuals. Importantly, just over half of these diseases have a known genetic cause. This leaves thousands of disease genes waiting to be discovered and millions of affected individuals without a diagnosis. The investigators will address these critical issues in genomic medicine by using genome sequencing and other 'omics technologies to assess patients whose comprehensive clinical workups have failed to yield a diagnosis. The hypothesis is that, when carefully selected, these undiagnosed disease patients will be a rich resource for new disease gene discovery.

This study is the research arm of the UW Undiagnosed Disease program (UW-UDP). The primary objective of this study is to discover new disease genes and expand the known phenotypes of rare Mendelian disorders. The secondary objectives are: a) Diagnose individuals with genetic disorders who have not been diagnosed using conventional clinical means and provide them with actionable knowledge to manage their disorders; b) Improve our understanding of the pathobiology of genetic disorders and the relationships between genomic variation and disease; and c) Develop and trial novel diagnostic technologies and analytics.

These objectives will be achieved through three aims:

Aim 1: Identify candidate disease variants in individuals suspected of an undiagnosed genetic disorder through the use of trio short read genome sequencing and data sharing with the rare disease databases GeneMatcher and MatchMaker Exchange.

Aim2: Further evaluate those individuals not diagnosed in Aim 1 by using novel 'omics technologies and bioinformatics algorithms. These approaches include a) ultra-long read de novo assembly-based genomic sequencing; b) RNA-Seq; c) epigenomics profiling, and d) conformational analysis of chromatin organization.

Aim 3: Provide functional assessments of selected candidate disease genes and genomic variants discovered in Aims 1 and 2 through collaborations with UW and external model organism researchers. These efforts will be facilitated through the use of a UW model organism researcher database that is linked to the Canadian Rare Diseases Models and Mechanisms Network database and an emerging global network of model organism researcher databases.

This research project is closely integrated with the UW-UDP's comprehensive clinical evaluations of undiagnosed patients. The standard clinical care component entails patient referral, collection and pre-visit assessment of medical records, and clinic visits for extensive phenotyping at the beginning of the study and for the return of results at the end of the study. The research workflow includes genome sequencing, data sharing with global disease gene discovery networks, and follow-up studies to determine causality of variants identified by genetic testing. This study will advance understanding of the pathobiology of genetic disease, improve clinical diagnostics, and aid in the diagnosis and management of individuals with previously undiagnosed rare disorders both within Wisconsin and beyond its borders.

ELIGIBILITY:
Inclusion Criteria:

* The applicant has a condition that remains undiagnosed despite thorough evaluation by healthcare providers (including clinical genetic testing).
* The applicant has at least one objective finding that is likely to have an identifiable genetic etiology.
* The applicant likely has a currently undescribed/new genetic condition or a known genetic condition associated with a novel gene.
* The applicant/legal guardian agrees to the collection, storage and recurrent sharing of coded information and biomaterials for research and diagnostic purposes both within and outside of the University of Wisconsin-Undiagnosed Diseases Program (UW-UDP)
* The applicant/legal guardian agrees to receive secondary findings from genetic testing.
* The applicant/legal guardian has sufficient proficiency in English to understand the consent.

Exclusion Criteria:

* The applicant already has a diagnosis that explains the objective findings.
* A specific diagnosis is suspected and a standard clinical workup performed by the referring/primary care provider would be appropriate.
* The UW-UDP is unlikely to improve on the comprehensive workup the applicant has already received.
* The applicant's symptoms are likely multifactorial or due to a non-genetic cause.

Max Age: 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Males and females, ages 0-100 years, of all races and ethnicities, with an undiagnosed disease despite thorough evaluation by healthcare providers and having at least one objective finding. Subjects can come from all states of the US, as well as from other countries.
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2021-07-16 (Actual); Primary Completion 2030-10 (Estimated); Study Completion 2030-10 (Estimated)

PRIMARY OUTCOMES:
Number of New Disease Genes Discovered | up to 5 years
Number of Expanded Disease Gene Phenotypes | up to 5 years

SECONDARY OUTCOMES:
Number of Participants who are Diagnosed in 5 years | up to 5 years
  A secondary objective of this study is to diagnose individuals with genetic disorders who have not been diagnosed using conventional clinical means and provide them with actionable knowledge to manage their disorders. This will be measured as the rate of diagnosis over the entire study.
Number of Participants Diagnosed per Analytical Technique | up to 5 years
  A secondary aim of this study is to develop and trial novel diagnostic technologies and analytics. The diagnosis rate per novel analytic technique will be assessed.
Diagnostic Rate by Disease Presentation | up to 5 years
  To improve understanding of the pathobiology of genetic disorders and the relationships between genomic variation and disease, number of participants diagnosed by disease presentation will be reported.

CONTACTS AND LOCATIONS:
Overall Officials: Bryn Webb, MD, Principal Investigator — University of Wisconsin, Madison
Locations (1):
- University of Wisconsin School of Medicine and Public Health, Madison, Wisconsin, United States

IPD SHARING:
Plan to Share IPD: Yes
Data from the UW-UDP will be shared via PhenomeCentral (https://www.phenomecentral.org) and Matchmaker Exchange (https://www.matchmakerexchange.org/).
  Data, images, and/or specimens will be shared in compliance with the NIH Genomic Data Sharing Policy and with other clinicians and researchers who may have similar patients and/or specific expertise/assays relevant to the participant's disorder. In this regard, a limited amount of non-PHI containing patient data will be shared with pre-vetted model organism collaborators at UW and elsewhere via our Center's local node of the Rare Diseases Models and Mechanisms Network (http://rdmmn.biotech.wisc.edu). This network facilitates the identification of model organism researchers who are willing and able to functionally assess the pathogenicity of candidate disease gene variants in rare disease patients (see http://www.rare-diseases-catalyst-network.ca for details).